CLINICAL TRIAL: NCT00933543
Title: A Double Blinded, Prospective, Randomized, Stratified, Placebo-controlled, Multi-center Study of Photodynamic Therapy With VisonacTM Cream in Patients With Moderate to Severe Acne Vulgaris.
Brief Title: Efficacy and Safety Study With Visonac Photodynamic Therapy (PDT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC TA204/09
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-11

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Moderate to severe
MeSH Terms: conditions — Acne Vulgaris | interventions — Red Light; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visonac cream with PDT (Experimental): Active treatment, Light dose 37 J/cm2.
  Interventions: Drug: Visonac PDT (MAL PDT); Procedure: PDT
- Vehicle cream with PDT (Placebo Comparator): Placebo treatment, Light dose 37 J/cm2.
  Interventions: Drug: Vehicle cream (placebo); Procedure: PDT

INTERVENTIONS:
Drug: Visonac PDT (MAL PDT) — Cream application followed by illumination with red light.
  Other Names: Visonac; MAL PDT; red light
  Arms: Visonac cream with PDT
Drug: Vehicle cream (placebo) — Cream application followed by illumination with red light.
  Other Names: Vehicle cream; MAL PDT; red light
  Arms: Vehicle cream with PDT
Procedure: PDT — Photodynamic Therapy - Light dose 37 J/cm2
  Other Names: Red light

SUMMARY:
The purpose of this trial is to study the efficacy and safety of Visonac PDT in patients from 9 to 35 years old with Aktilite® CL512. Patients was randomized to Visonac or vehicle cream without occlusion and red light(dose: 37J/cm2)

DETAILED DESCRIPTION:
Double blinded, prospective, randomized, stratified, placebo-controlled, multi-center study in patients with moderate to severe acne vulgaris. Patients with facial severity grades 3 to 4 on the Investigator's Global Assessment (IGA) scale will be included. Each patient will be classified according to age in the two age groups 9 to 12 years and 13 to 35 years and randomized to either Visonac or vehicle cream within each age group. All patients will receive 4 treatments 2 weeks apart (at week 0, 2 ,4 and 6 week). Efficacy evaluation will be done after each treatment and at 12 weeks after the first treatment. Safety evaluations will be performed at each treatment visit and at 12 weeks after the first treatment.

Photographs of patients will be taken before and after treatment at first and last treatment visit, and at 12 weeks after first treatment.

Blood samples will be drawn at 3 visits; pre-treatment visit, one week after first treatment and at one week after last treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients, above 9 years of age with moderate to severe facial acne vulgaris (IGA score 3-4).
* Female patients who are surgically sterile, pre-menstrual, postmenopausal, abstinent, or willing to use an adequate means of contraception including birth control pills, or barrier methods and spermicide for at least 14 days prior to T1. Patients using birth control pills must have used the same product and dose for at least 6 months and must agree to stay with the same product and dose for an additional 6 months.
* Fitzpatrick skin type I through VI.
* Patients with 20 to 100 inflammatory lesions (papules, pustules, and nodules) on the face.
* Patients with 30 to 120 non-inflammatory lesions (open and closed comedones) on the face.
* Patients with no more than 2 nodular lesions on the face.
* Signed and verified informed consent form. For subjects under age of 18, an assent form in conjunction with an informed consent form, signed and verified by parent/guardian.

Exclusion Criteria:

Patients presenting with any of the following will not be included in the study:

* Patient is the investigator or any sub investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* Patients unlikely to comply with the protocol, e.g., mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the clinical study, uncooperative attitude or unlikelihood of completing the study (e.g., drug or alcohol abuse).
* Female patients using oral contraceptives, that have not used the same product or dose within the last 6 months and do not agree to stay with the same product and dose for the duration of the study.
* Pregnancy
* Patients undergoing testosterone or any other systemic hormonal treatment.
* Patients using hormonal contraceptives solely for the control of acne.
* Known allergy to MAL, to a similar PDT compound, or to excipients of the cream.
* Patients with porphyria.
* Patients with cutaneous photosensitivity.
* Participation in other clinical studies either concurrently or within the last 30 days, before T1.
* Patients with a washout period for topical treatments e.g., topical BPOs, retinoids and antibiotics, for their acne of less than 14 days, before T1. Medicated cleansers may be used during the washout period and stopped before the treatment.
* Patients with a washout period for oral antibiotics for treatment of their acne of less than 1 month, before T1.
* Patients with a washout period for oral isotretinoin of less than 6 months, before T1.
* Patients with a beard or other facial hair that might interfere with study assessments.
* Patients with melanoma or dysplastic nevi in the treatment area.
* Exposure to ultraviolet radiation (UVB phototherapy, sun tanning salons) within the last 30 days.
* Exposure to PDT within 12 weeks before T1.

Ages: 9 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence F. Eichenfield, M.D, Principal Investigator — Children's Specialists of San Diego / Rady Children's Hospital San Diego
Locations (11):
- United States (8):
  - Children's Specialists of San Diego / Rady Children's Hospital San Diego, San Diego, California
  - DeNova Research, Chicago, Illinois
  - Dermatology Institute of DuPage Medical Group, Naperville, Illinois
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Dermatology Associates of Rochester, Rochester, New York
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Madison Skin & Research, Inc, Madison, Wisconsin
- Canada (3):
  - Windsor Clinical Research, Inc., Windsor, Ontario N8W 5L7, Ontario
  - INNOVADERM Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from September-December 2009. Dermatology clinics, with pediatric patients
Period: Overall Study
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Started | 54 | 53
Completed | 51 | 46
Not Completed | 3 | 7
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lack of Efficacy | 0 | 3
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT | Total
Number analyzed (Participants) | 54 | 53 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 34 | 69
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 27 | 59
  Male | 22 | 26 | 48
Region of Enrollment [Number; unit: participants]
  Canada | 17 | 16 | 33
  United States | 37 | 37 | 74
Patients with mild and moderate hyperpigmentation [Number; unit: number of patients]
  No hyperpigmentation | 39 | 34 | 73
  Mild hyperpigmentation | 5 | 10 | 15
  Moderate hyperpigmentation | 8 | 8 | 16
  Severe hyperpigmentation | 2 | 1 | 3
Investigator Global Assessment (IGA) Score [Number; unit: participants]
  IGA 3 (Moderate acne) | 44 | 45 | 89
  IGA 4 (Severe acne) | 10 | 8 | 18
Fitzpatrick Skin type [Number; unit: participants] — I: White; very fair; red or blond hair; blue eyes; freckles Always burns, never tans II: White; fair; red or blond hair; blue, hazel or green eyes Usually burns, tans with difficulty III: Cream white; fair with any eye or hair color; very common Sometimes mild burn, gradually tans IV: Brown; typical Mediterranean Caucasian skin Rarely burns, tans with ease V: Dark brown; Middle Eastern skin types Very rarely burns, tans very easily VI: Black Never burns, tans very easily
  participants
    Skin type I | 5 | 6 | 11
    Skin type II | 14 | 15 | 29
    Skin type III | 24 | 21 | 45
    Skin type IV | 4 | 6 | 10
    Skin type V | 5 | 2 | 7
    Skin type VI | 2 | 3 | 5
Scarring [Number; unit: number of patients] — The investigator assess the scarring using a scale called SCAR-S. Clear 0: No visible scars from acne. Almost clear 1: Hardly visible scars from 2.5 meters away. Mild 2: Easily recognizable, less than ½ the affected area (eg. face, back or chest) involved.
  Moderate 3: More than ½ affected area (eg. face, back or chest) involved. Severe 4: Entire area involved. Very severe 5: Entire area with prominent atrophic or hypertrophic scars.
  number of patients
    Patients with no scarring | 21 | 26 | 47
    Patients with almost clear scarring | 9 | 10 | 19
    Patients with mild scarring | 15 | 9 | 24
    Patients with moderate scarring | 6 | 6 | 12
    Patients with severe scarring | 3 | 1 | 4
    Patients with very severe scarring | 0 | 1 | 1
Patients with dryness [Number; unit: Number of patients] — The investigator assess the dryness using a scale from 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe).
  Number of patients
    No dryness | 45 | 46 | 91
    Mild dryness | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Success According to the Dichotomized IGA Scale Based on Facial Assessments 12 Weeks After the First Treatment. Success is Defined as an Improvement of at Least 2 Grades From the Baseline Score.
Time Frame: 12 weeks after the first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 53
percentage of participants | 9.26 [1.53 to 16.99] | 1.89 [0.00 to 5.55]
Statistical Analysis 1: Comparison: Visonac Cream With PDT vs Vehicle Cream With PDT; H0: τ (Vehicle PDT) = τ (MAL PDT) versus HA: τ (Vehicle PDT) ≠ τ (MAL PDT); Test type: Superiority or Other; p = 0.0703, Cochran-Mantel-Haenszel — Priori threshold for statistical significance was 5%; Cochran-Mantel-Haenszel (CMH) test stratified by center. No adjustment for multiple comparisons was done; Odds Ratio (OR) = 6.43, 95% CI 2-sided [0.65 to 63.18]

2. Secondary Outcome: Percent Change From Baseline in Facial Inflammatory (Nodules, Papules, and Pustules)Lesion Count
Time Frame: 6 weeks after the first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 53
percent change from baseline | -35.4 (30.85) | -20.3 (38.72)

3. Primary Outcome: Absolute Change From Baseline in Facial Inflammatory Lesion Count (Nodules, Papules, and Pustules)
Time Frame: 12 weeks after the first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 53
lesions | -14.0 (17.94) | -13.8 (23.76)
Statistical Analysis 1: Comparison: Visonac Cream With PDT vs Vehicle Cream With PDT; H0: τ (Vehicle PDT) = τ (MAL PDT) versus HA: τ (Vehicle PDT) ≠ τ (MAL PDT); Test type: Superiority or Other; p = 0.2969, ANCOVA — Priori threshold for statistical significance was 5%; ANCOVA model, including center and baseline lesion count as a covariates; Mean Difference (Net) = -3.92, 95% CI 2-sided [-11.35 to 3.50]

4. Primary Outcome: Absolute Change From Baseline in Facial Non Inflammatory Lesion Count
Time Frame: 12 weeks after first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 53
lesions | -14.3 (26.54) | -17.1 (25.84)
Statistical Analysis 1: Comparison: Visonac Cream With PDT vs Vehicle Cream With PDT; H0: τ (Vehicle PDT) = τ (MAL PDT) versus HA: τ (Vehicle PDT) ≠ τ (MAL PDT); Test type: Superiority or Other; p = 0.8913, ANCOVA — Priori threshold for statistical significance was 5%; ANCOVA model, including center and baseline lesion count as a covariates; Mean Difference (Net) = 0.67, 95% CI 2-sided [-9.09 to 10.43]

5. Secondary Outcome: Percent Change From Baseline in Facial Inflammatory (Nodules, Papules, and Pustules)Lesion Count
Time Frame: 12 weeks after the first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 53
Percent change from baseline | -33.1 (39.34) | -27.5 (44.38)

6. Secondary Outcome: Percent Change From Baseline in Facial Non Inflammatory Lesion Count
Time Frame: 6 weeks after first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 53
percentage change from baseline | -25.3 (39.72) | -15.8 (47.11)

7. Secondary Outcome: Percent Change From Baseline in Facial Non Inflammatory Lesion Count
Time Frame: 12 weeks after first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 53
percentage change from baseline | -26.0 (52.23) | -24.4 (37.66)

8. Secondary Outcome: Percent Change From Baseline in Facial Total Lesion Count
Time Frame: 6 weeks after the first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 52 | 52
Percent change from baseline | -29.5 (27.72) | -18.0 (35.39)

9. Secondary Outcome: Percent Change From Baseline in Facial Total Lesion Count
Time Frame: 12 weeks after the first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 53
Percent change from baseline | -29.8 (36.04) | -26.8 (29.61)

10. Secondary Outcome: Proportion of Patients With a Reduction of at Least 50% From Baseline in Facial Non-inflammatory Lesion Count
Time Frame: 12 weeks after last treatment
Population: ITT
Measure: Number; unit: participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 53
participants | 17 | 10

11. Secondary Outcome: Proportion of Patients With a Reduction of at Least 50% From Baseline in Facial Inflammatory Lesion Count From Baseline
Time Frame: 12 weeks after first treatment
Measure: Number; unit: participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 53
participants | 20 | 19

12. Secondary Outcome: Absolute Change From Baseline in Facial Inflammatory Lesion Count
Time Frame: 6 weeks after the first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 52 | 52
lesions | -17.5 (9.0) | -10.8 (22.41)

13. Secondary Outcome: Absolute Change From Baseline in Facial Non- Inflammatory Lesion Count
Time Frame: 6 weeks after the first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 52 | 52
lesions | 12.9 (21.41) | 11.3 (28.24)

14. Secondary Outcome: Absolute Change From Baseline in Facial Total Lesion Count
Time Frame: 6 weeks after the first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 52 | 52
lesions | -27.2 (26.19) | -20.6 (36.68)

15. Secondary Outcome: Proportion of Patients With Success According to the Dichotomized IGA Scale Based on Facial Assessments 12 Weeks After the First Treatment. Success is Defined as an Improvement of at Least 2 Grades From the Baseline Score.
Time Frame: 6 weeks after the first treatment
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 52 | 52
Participants | 3 | 1

16. Secondary Outcome: Facial Pain Assessed Using a Visual Analogue Scale From 0 to 10, Where 0 Indicates no Pain and 10 Indicates Worst Pain Imaginable
Description: Facial pain was assessed on a visual analogue scale ranging from 0-10cm.
Time Frame: directly after first treatment
Population: Safety population
Measure: Mean (Full Range); unit: cm
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 53
cm | 1.5 (2.2) [0.0 to 9.8] | 0.28 (0.64) [0.0 to 3.6]

17. Secondary Outcome: Facial Pain Assessed Using a Visual Analogue Scale From 0 to 10, Where 0 Indicates no Pain and 10 Indicates Worst Pain Imaginable
Description: Facial pain was assessed on a visual analogue scale ranging from 0-10cm.
Time Frame: directly after second treatment
Population: Safety population
Measure: Mean (Full Range); unit: cm
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 52 | 52
cm | 1.37 [0.0 to 8.5] | 0.15 [0.0 to 1.6]

18. Secondary Outcome: Facial Pain Assessed Using a Visual Analogue Scale From 0 to 10, Where 0 Indicates no Pain and 10 Indicates Worst Pain Imaginable
Description: Facial pain was assessed on a visual analogue scale ranging from 0-10cm.
Time Frame: directly after third treatment
Population: Safety population
Measure: Mean (Full Range); unit: cm
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 51 | 50
cm | 1.53 [0.0 to 8.1] | 0.17 [0.0 to 1.4]

19. Secondary Outcome: Facial Pain Assessed Using a Visual Analogue Scale From 0 to 10, Where 0 Indicates no Pain and 10 Indicates Worst Pain Imaginable
Description: Facial pain was assessed on a visual analogue scale ranging from 0-10cm.
Time Frame: directly after fourth treatment
Population: Safety population
Measure: Mean (Full Range); unit: cm
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 51 | 49
cm | 1.39 [0.0 to 8.2] | 0.19 [0.0 to 2.6]

20. Secondary Outcome: Proportion of Patients With Mild and Moderate Hyperpigmentation
Time Frame: at 12 weeks after first treatment
Population: Safety
Measure: Number; unit: participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 49
participants | 26 | 32

21. Secondary Outcome: Proportion of Patients With Severe Hyperpigmentation
Time Frame: at 12 weeks after first treatment
Population: Safety
Measure: Number; unit: participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 49
participants | 1 | 0

22. Secondary Outcome: Proportion of Patients With Mild or Moderate Scarring at End of Study
Time Frame: week 12
Measure: Number; unit: participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 49
participants | 36 | 34

23. Secondary Outcome: Proportion of Patients With Clear or Almost Clear Scarring at End of Study
Time Frame: week 12
Measure: Number; unit: participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 49
participants | 59 | 63

24. Secondary Outcome: Proportion of Patients With Severe and Very Severe Scarring at End of Study
Time Frame: week 12
Measure: Number; unit: participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 49
participants | 6 | 2

25. Secondary Outcome: Proportion of Patients With Hypopigmentation (Mild Moderate, Severe)
Time Frame: at 12 weeks after first treatment
Population: Safety
Measure: Number; unit: participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 49
participants | 0 | 0

26. Secondary Outcome: Proportion of Patients With Dryness (Mild)
Time Frame: at 12 weeks after first treatment
Population: Safety
Measure: Number; unit: participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 54 | 49
participants | 20 | 16

ADVERSE EVENTS:
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/53
Other Adverse Events (participants affected / at risk) | 46/54 | 32/53
OTHER ADVERSE EVENTS (reported when occurring in more than 2.8% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Visonac Cream With PDT (N=54) | Vehicle Cream With PDT (N=53)
Erythema (Skin and subcutaneous tissue disorders) | 26 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 8
Skin burning sensation (Skin and subcutaneous tissue disorders) | 12 | 4
Skin irritation (Skin and subcutaneous tissue disorders) | 4 | 0
Pain (General disorders) | 27 | 6
Facial pain (General disorders) | 4 | 4
Feeling hot (General disorders) | 2 | 2
Nasopharyngitis (Infections and infestations) | 10 | 5
Paraestehesia (Nervous system disorders) | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days